CLINICAL TRIAL: NCT07154914
Title: Mapping Prostate Cancer Evolution and Therapy Resistance With Single-Cell Technologies
Brief Title: A Novel Insight Into CRPC Progression and Immune: Evidence From Single-cell Spatial Transcriptome Multi-omics
Status: Not yet recruiting | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Dr. Zhang Meng, Prof., Anhui Medical University
Other Study IDs: AYFY2025-08-27
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cance
MeSH Terms: interventions — abiraterone; Androgen Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Abiraterone + ADT — Patients receiving androgen deprivation therapy (ADT) combined with abiraterone. Abiraterone is a CYP17A1 inhibitor used in combination with prednisone and ADT for metastatic hormone-sensitive prostate cancer (mHSPC). This combination is given in real-world practice according to clinical guidelines.

SUMMARY:
This study will follow patients with metastatic hormone-sensitive prostate cancer (mHSPC) who receive androgen deprivation therapy (ADT) combined with different treatments. Prostate cancer is a common cancer in men, and many patients in China are diagnosed at an advanced stage. While ADT alone has been the standard treatment, most patients eventually progress to castration-resistant disease.

New medicines such as abiraterone, enzalutamide, apalutamide, darolutamide, and chemotherapy like docetaxel have shown survival benefits when added to ADT. This study aims to observe how different ADT-based combinations work in real-world practice and whether genetic differences affect outcomes.

About 396 patients will be enrolled and followed until disease progression or death. The results will help identify which treatments are most effective and guide more personalized care for men with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients, age >18 and <85 years.
2. Histologically confirmed prostate adenocarcinoma, ductal adenocarcinoma, or intraductal carcinoma.
3. Evidence of distant metastases by imaging (according to RECIST criteria).
4. No prior systemic therapy for prostate cancer (no ADT or other systemic treatments).
5. ECOG performance status 0-2 and estimated life expectancy >6 months.
6. Adequate organ function as indicated by:

   * Hemoglobin ≥ 90 g/L

     * ANC ≥ 1.5 × 10^9/L

       * Platelet count ≥ 75 × 10^9/L

         * WBC ≥ 3 × 10^9/L ⑤ Total bilirubin ≤ ULN ⑥ ALT/AST ≤ 2.5 × ULN ⑦ Creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula)

           * INR ≤ 1.5 or PT < 4 sec above ULN
7. Ability to provide written informed consent.

Exclusion Criteria:

1. Histological diagnosis of neuroendocrine or small-cell prostate cancer.
2. No evidence of distant metastases on imaging.
3. Prior systemic therapy for prostate cancer (neoadjuvant, adjuvant, or systemic).
4. Severe endocrine, metabolic, gastrointestinal, hepatic, or renal disease (including chronic hepatitis, cirrhosis, chronic nephritis, or renal failure).
5. History of immunodeficiency, including HIV positivity, congenital immunodeficiency, or organ transplantation.
6. History of other malignancies (except non-melanoma skin cancer).
7. Concurrent participation in another clinical trial.
8. Inability to provide clinical information or anticipated loss to follow-up.
9. Any condition deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 85 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Male patients with newly diagnosed metastatic hormone-sensitive prostate cancer (mHSPC), recruited from multiple centers in China. Eligible patients are treatment-naïve and will receive androgen deprivation therapy (ADT) combined with different regimens according to real-world clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to progression to castration-resistant prostate cancer (CRPC) | Up to 36 months